CLINICAL TRIAL: NCT04721795
Title: Repurposing a Lipid Lowering Drug to Treat Tuberculosis: Effectiveness of Statins as Adjuvant to Treatment of Pulmonary Tuberculosis in Nigeria
Brief Title: Treating Tuberculosis With the Lipid Lowering Drug Atorvastatin in Nigeria(ATORvastatin in Pulmonary TUBerculosis)
Acronym: ATORTUB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Cures Within Reach (Other)
Responsible Party: Principal Investigator, Adewole Olufemi, Principal Investigator/Consultant Physician and Professor of Medicine, Obafemi Awolowo University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERC/2020/10/05; NHREC/27/02/2009a (Other: NHREC)
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis
Keywords: lipids drugs; atorvastatin; outcome
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Rifampin; Isoniazid; Pyrazinamide

STUDY DESIGN:
Intervention Model Description: Randomised
Who Masked: Outcomes Assessor
Masking Description: Outcome assesor is blinded to treatment groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin with standard anti tuberculosis drugs (Experimental): Participants will receive oral 30/40mg of atorvastatin daily for 2 months together with oral doses of standard antituberculosis drugs consisting of Rifampicin, INH, Ethambuthol and pyrazinamide for 2months. At the end of 2months, participants will continue with only standard anti tuberculosis drugs, Rifampicin and INH for 4months.Doseage of antituberculosis drugs are dependent on weight
  Interventions: Drug: Atorvastatin with standard anti tuberculosis drugs
- Anti tuberculosis drugs only (Active Comparator): Participants will receive oral doses of standard antituberculosis drugs only consisting of Rifampicin, INH, Ethambuthol and pyrazinamide for 2months. At the end of 2months, participants will continue with only standard anti tuberculosis drugs, Rifampicin and INH for 4months.Doseage of antituberculosis drugs are dependent on weight
  Interventions: Drug: Standard anti tuberculosis drugs only

INTERVENTIONS:
Drug: Atorvastatin with standard anti tuberculosis drugs — Participants will receive oral 30/40mg of atorvastatin daily for 2 months together with oral doses of standard antituberculosis drugs consisting of Rifampicin, INH, Ethambuthol and pyrazinamide for 2months. At the end of 2months, participants will continue with only standard anti tuberculosis drugs, Rifampicin and INH for 4months.Doseage of antituberculosis drugs are dependent on weight
  Other Names: Atorvastatin, Statins
  Arms: Atorvastatin with standard anti tuberculosis drugs
Drug: Standard anti tuberculosis drugs only — Participants will receive oral doses of standard antituberculosis drugs consisting of Rifampicin, INH, Ethambuthol and pyrazinamide for 2months. At the end of 2months, participants will continue with only standard anti tuberculosis drugs, Rifampicin and INH for 4months.Doseage of antituberculosis drugs are dependent on weight
  Other Names: Rifampicin, INH, Ethambuthol and Pyrazinamide
  Arms: Anti tuberculosis drugs only

SUMMARY:
Tuberculosis (TB) is caused by mycobacterial organism. It is the leading infectious disease cause of death globally, with more than 10 million new cases and over 2 million deaths annually. Developing countries bear the greatest brunt of the disease. The long duration of current treatment is associated with poor compliance, thereby contributing to frequent relapses and to the emergence of drug-resistant TB. In addition, individuals who have been clinically cured may have lung damage, which could be permanent. Therefore, new and more effective therapeutic agents against TB are needed. Emerging evidence has shown that lipid lowering drugs like statins can make the TB bacteria more susceptible to current treatments. This proof-of-concept clinical trial will add the repurposed drug atorvastatin, commonly used to reduce cholesterol levels, to the standard therapies of TB patients in Nigeria. Atorvastatin is a well-tolerated and safe drug, and its addition is expected to accelerate clearance of the TB-causing bacteria without additional side effects. If this research is successful, it could provide evidence for using a common, easily available generic drug to improve treatment of one of the most debilitating infectious diseases.

DETAILED DESCRIPTION:
INTRODUCTION Tuberculosis is a chronic disease responsible for most deaths from infectious disease with an estimated I0 million cases and close to 2million deaths globally. 1 Despite the availability of therapy for TB, the scourge of the disease has not abated especially in the developing countries. The disease is caused by a bacterium called Mycobacterium tuberculosis, a non-spore forming intracellular organism. TB exists in two forms; primary and secondary infection. While primary infection most times goes unnoticed and are usually associated with non-specific symptoms, secondary infections are usually associated with profound symptoms and signs in various organs especially in the lungs. Majority of persons overcome primary infection but the tubercule bacilli may lie dormant in the macrophages.2 Secondary infection occurs as a result of either endogenous reactivation or exogenous re-infection. Pulmonary TB is responsible for more than 85% of the cases.

MTB infect and survive humans by evading the various immune defense systems.3 The organism accumulates and utilizes an abundant amount of lipids and cholesterol for its cell wall, and as a source of carbon for synthesis of virulence factors. 4 Mycobacterium tuberculosis also utilizes cholesterol as a vehicle to enter macrophage, inhibit phagocytosis and inhibit growth and development of phagocytes.5 These greatly impairs the hydrolytic and antimicrobial properties and activities of phagocytes.5,6 Current therapy is as old as the disease itself; is of long duration, hence it is associated with poor compliance. This contributes to frequent relapses and emergence of resistant form of the disease. Average interval between one episode of TB and another range from 6-18 months after completion of therapy. Despite clinical cure, approximately half of patients have permanent lung damage. In Nigeria, TB is a major risk factor for Chronic Obstructive Pulmonary Disease, lung fibrosis/scarring and other diseases. It is clear that new and innovative therapeutic agents are needed to tackle this hydra- headed disease. In order to address these challenges, a lipid lowering agent, atorvastatin is being repurposed.

The use of statins have been demonstrated in infectious diseases and especially in tuberculosis than other organisms.7 In vitro studies have demonstrated that statins could strengthen the host response against M. tuberculosis and inhibit the activation of T cells induced by M. tuberculosis antigens.8,9 In another study, murine bone marrow-derived macrophages that were exposed to simvastatin and were infected with M. tuberculosis, showed a significant reduction in mycobacterial growth, without adverse effects on cell viability.10 Treatment of TB in animal model with statins and anti TB drugs showed that treatment with anti-TB drugs plus simvastatin reduced the percentage of relapses by 50% compared with treatment with only anti-TB drugs.11 Taken together, all these studies in animal model indicate that statins has anti-TB effect, reduces bacillary load, shortens the duration of therapy and decreases relapse rate when used with first-line anti-TB drugs.

Most of the clinical evidence on the role of statins in TB were from retrospective and nested case control studies from Asian continent.12,13 In one study in Taiwan, diabetic subjects older than 65 treated with statins had a lower risk of developing active tuberculosis, with a risk of 0.76 (95% CI, 0.60-0.97). 12 Chronic use of statins (more than 90 days) was associated with the lowest risk (RR 0.62; 95% CI 0.53-0.72) as shown in another study.13 Within the limits of the designs of these studies, the positive and protective role of statins in TB in humans were demonstrated and has provided basis for further studies. This proposal seeks to provide robust evidence in a well designed study, for repurposing statins to treat TB.

If this is successful, the investigators anticipate a significant improvement in health and well being for patients. Patients will have the option of being treated with an effective and safe regimen with minimal side effects including patients with HIV/TB co-infection, as statins can be co-administered safely with antiretroviral drugs. Additionally, the investigators anticipate a reduction in relapse rate, persistence and resistance to Mycobacterium tuberculosis. Currently, patients still experience post treatment non-infectious complications that limit their functionality. The investigators anticipate this treatment will mitigate against this and lead to improvement in the quality of life of patients and survivors. Both direct and indirect costs of the disease can be rechanneled to revamp the health system and other economic potentials of the developing world. If this prove successful, there would be an accelerated and significant progress to achieving the World Health Organization and End TB Sustainable Development Goals. Overall the investigators anticipate a great turn around in the socio-economic life of people and countries of the developing world where TB has caused untoward and unimaginable stagnation.

1.3 Study Design

Experimental design/Research Plan The investigators propose a Phase IIA/IIB randomized open label trial to evaluate the safety, tolerability, pharmacokinetics(PK), and efficacy of atorvastatin in subjects with uncomplicated, smear-positive, drug-susceptible pulmonary tuberculosis. See Figure I.

Consented and eligible patients with active tuberculosis will be recruited and be randomized to receive either 30/40mg of atorvastatin with standards anti-TB drugs for 2months or the standards anti-TB drugs alone for 2months. Randomization will be based on Zelen rule 14 and follow a predefined allocation ratio of 1:1

Phase IIA will seek to determine the safety and early bactericidal efficacy of atorvastatin in combination with standard anti-TB in 40 patients. Phase IIB, will seek to determine safety, and sputum culture conversion of atorvastatin in combination with standard anti-TB compared with standard anti-TB drugs alone after 2months in a total of 150 patients. Figure I.

Patients will be hospitalized for supervised drug administration and assessed daily for vital signs and adverse effects AEs especially at phase IIA. Semi intensive profiling of plasma atorvastatin concentrations with a validated high-performance liquid chromatography will be conducted after the first dose on day 1 through to the last dose on day 14. Sputum will be collected for 16hours overnight for two nights before drug intake, daily from days 1 to 4, and every alternate day until day 14 in both cohorts. Samples will be transported and refrigerated till colony forming unit is done. Full blood count, coagulation studies, serum chemistry, lipid profile, Creatinine phosphokinase, urinalysis, and 12-lead electrocardiograms (ECGs) will be performed prior to drug intake and at regular intervals during and at 2 weeks. Patients recruited for this phase will continue in the assigned study arm and join the phase IIB.

Interim analysis will be done in the two groups at the end of the 2weeks with particular emphasis on safety profile, incidence and number of adverse effects, bactericidal activity and a preliminary report of serum levels of atorvastatin in two groups.

For the phase IIB, patients will be randomized as previously stated into any of the two groups and will be monitored closely. Sputum will be collected at 4, 6 and 8 weeks for smear/GenXpert. At the end of 8 weeks, sputum will be collected overnight for MTB culture in addition. During this period, number and types of AEs in the participants will also be noted. At the end, patients will be discharged from the study to continue and complete course of standard anti-tuberculosis chemotherapy. To determine the performance of the Sweat TB test, patients will be prospectively enrolled and the results from the test compared with sputum/GenXpert result.

All investigations will be done at laboratories at OAU/OUATHC, Ile Ife. Microbiological assessment including CFU/ culture conversion will be done at the Mycobacterial Laboratory, OAU/OAUTHC, Ile Ife. Drug assays will be done at the collaborating center; Birmingham Heartlands Hospital/University of Birmingham, UK

Patients will not be coerced to enroll in the study but they will be allowed to enroll after full written and informed consent. However they will be encouraged to attend all clinic and research appointment. However in order to ensure adherence to research protocol especially the period they need to be assessed, they will be provided with transport fare for the period of evaluation. For the initial 2 weeks of hospilisation, all fee including feeding will be borne by the research.

.

2.0 STUDY OBJECTIVES B. SPECIFIC AIMS, EXPECTED MEASURABLE OUTCOMES AND DELIVERABLES.

1.1.Specific aims:

1. To determine the safety profile of atorvastatin in combination with anti-TB drugs
2. Determine the efficacy of atorvastatin in treating patients with tuberculosis, i.e if atorvastatin has early bactericidal activity and effect on sputum culture conversion
3. To determine the pharmacodynamics and pharmacokinetics of atorvastatin in combination with anti-TB drugs in patients with active TB

1.2. Primary outcome measures:

1. Efficacy of atorvastatin treatment in combination with standard anti-TB chemotherapy as measured by:

   1. Sputum conversion at 2 month as measured by the number of patients with a negative culture at 2 months
   2. Time to sputum conversion as measured by the time interval to the first sputum negative result with sputum smear microscopy/GenXpert [ Time Frame: up to 2 months
   3. Early Bactericidal Activity /Overall response rate associated with atorvastatin treatment in combination with standard anti-TB chemotherapy. [ Time Frame: up to 2weeks ) Measured as the Daily Rate of Change in log10 Colony Forming Units of M. Tuberculosis in Sputum on Solid Media [ Time Frame: up to 2weeks )
2. Incidence of treatment-emergent adverse events associated with atorvastatin treatment in combination with standard anti TB chemotherapy. [ Time Frame: up to 2 months ] The incidence of AEs will measured by the incidence of abnormalities in clinical laboratory tests (serum chemistry, hematology, urinalysis, and coagulation), physical examinations, vital signs, and electrocardiograms.

1.3. Secondary Outcome Measure :

1. Plasma level of atorvastatin in combination with standard anti TB chemotherapy [ Time Frame: up to 2 months ] Measured by Pharmacokinetics: Maximum Plasma Concentration (Cmax) of atorvastatin
2. Early bactericidal activity as measured by change in CFU for days 0-2 and 7-14

1.4. Exploratory Outcome measure:

1. Diagnostic utility of Sweat TB test in detecting tuberculosis. This is as measured by sensitivity, specificity, PPV and degree of agreement.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Newly diagnosed, uncomplicated, drug-susceptible pulmonary TB
  2. Sputum Smear, culture or GenXpert result positive for pulmonary TB
  3. Ability to provide written, informed consent prior to trial initiation
  4. Male or and non pregnant female participants between 18 and 65 years of age
  5. Body mass index 16.0 and 32.0 kg/m2
  6. Ability to produce an adequate volume of sputum (approximately 10 -15mL or more estimated overnight production).

     Exclusion Criteria:

     Exclusion Criteria:

  <!-- -->

  1. Participants known or suspected of having any form of drug resistance TB.
  2. Patients co infected with HIV
  3. Those with poor general condition where no delay in treatment can be tolerated
  4. Evidence of clinically significant metabolic or co morbid medical conditions ; malignancy; or other diseases like history of or current cardiovascular disorder such as heart failure, coronary heart disease, arrhythmia.
  5. Known or family history of bleeding disorders.
  6. Any renal impairment characterized by serum creatinine clearance of 1.5 x upper limit of normal of the clinical laboratory reference range at screening.
  7. Myositis and or Creatinine phosphokinase three times upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures Efficacy of atorvastatin treatment in combination with standard anti-TB chemotherapy | 2 months
  Sputum conversion at 2 month as measured by the number of patients with a negative culture
Time to sputum conversion | up to 2months
  Time to sputum conversion as measured by the time interval to the first sputum negative result with sputum smear microscopy/GenXpert
Early Bactericidal Activity | up to 2 weeks
  Overall response rate associated with atorvastatin treatment in combination Measured as the Daily Rate of Change in log10 Colony Forming Units of M. Tuberculosis in Sputum on Solid Media Overall response rate associated with atorvastatin treatment in combination with standard anti-TB chemotherapy
Incidence of treatment-emergent adverse events | Up till 2months
  Incidence of treatment-emergent adverse events associated with atorvastatin treatment in combination with standard anti TB chemotherapy.

SECONDARY OUTCOMES:
Plasma level of atorvastatin in combination with standard anti TB chemotherapy | Up to 2months
  Plasma level of atorvastatin in combination with standard anti TB chemotherapy

OTHER OUTCOMES:
Exploratory Outcome measure | up to 2months
  Diagnostic utility of Sweat TB test in detecting tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Olanisun P Adewole, MD, Principal Investigator — Obafemi Awolowo University Teaching Hospitals Complex; Bolanle A Omotoso, MD, Study Director — Obafemi Awolowo University Teaching Hospitals Complex
Locations (2):
- Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Osun State, Nigeria
- Birmingham Heartlands Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No